CLINICAL TRIAL: NCT03287115
Title: Biomarkers of Broccoli Intake: A Pilot Study to Characterize Novel Metabolites by Targeted Metabolic Profiling and Non-Targeted Metabolomics
Brief Title: Biomarkers of Broccoli Intake: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Craig Charron, Research Molecular Biologist, USDA Beltsville Human Nutrition Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS58
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Broccoli (Experimental): Subjects will consume a dose of broccoli on day 11
  Interventions: Other: Broccoli consumption

INTERVENTIONS:
Other: Broccoli consumption — All subjects will eat broccoli on day 11

SUMMARY:
The objectives of the study are 1) to characterize plasma and urinary metabolites that originate from glucobrassicin, 1-methoxyglucobrassicin, 4-methoxyglucobrassicin, and 4-hydroxyglucobrassicin, which are the major indole glucosinolates found in broccoli, and 2) to identify novel plasma and urinary metabolites following broccoli consumption that may have roles in reducing the risk of cancer.

DETAILED DESCRIPTION:
Consumption of Brassica vegetables is inversely associated with incidence of several cancers, including cancer of the lung, stomach, liver, colon, rectum, breast, endometrium, and ovaries. Brassicas are a good source of many nutrients, but the unique characteristic of Brassicas is their rich content of glucosinolates. Breakdown products of indole glucosinolates in Brassica vegetables show promise for reducing the risk of cancer, but have received comparatively less research attention than those of aliphatic glucosinolates. The aim of this study is to investigate plasma and urinary metabolites of indole glucosinolates from broccoli and to identify novel metabolites that may have roles in reducing cancer risk.

ELIGIBILITY:
Inclusion Criteria:

* Non tobacco user
* Cancer Free
* Not currently taking glucosinolate/isothiocyanate containing supplements

Exclusion Criteria:

* Type 2 diabetes requiring the use of diabetes pills, insulin, or non-insulin shots
* Use of blood-thinning medications such as Coumadin (warfarin), Dicumarol, or Miradon (anisindione)
* History of bariatric surgery or nutrient malabsorption disease (such as celiac disease) or other metabolic disorders requiring special diet recommendations
* Pregnant, lactating, or intending to become pregnant during the study period
* Crohn's disease or diverticulitis
* Suspected or known strictures, fistulas or physiological/mechanical GI obstruction
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
The change in glucosinolate metabolites will be measured in blood plasma and urine. | On Day 11
  To track the changes of indole glucosinolate metabolites, glucosinolate metabolites will be measured in both blood plasma and urine.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No